CLINICAL TRIAL: NCT05789537
Title: A Global, Open-label Study to Investigate the Efficacy and Safety of SerpinPC in Subjects with Hemophilia B with Inhibitors
Brief Title: A Study of SerpinPC in Participants with Hemophilia B (HemB) with Inhibitors
Acronym: PRESent-3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to business and strategic decision
Sponsor: ApcinteX Ltd (Industry)
Collaborators: Centessa Pharmaceuticals plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP-0103; 2022-502881-25-00 (Other: EU CT Number)
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hemophilia B with Inhibitor; Hemophilia B
Keywords: SerpinPC; Hemophilia
MeSH Terms: conditions — Hemophilia B; Hemophilia A | interventions — Protein C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SerpinPC (Experimental): Participants will receive SerpinPC 1.2 milligrams/kilogram (mg/kg) subcutaneous (SC) injection every 2 weeks (Q2W) for 48 weeks after a prospective observation of 12 weeks for all participants, either in a prior non-interventional study (AP-0105[NCT05605678]) or as part of the ongoing study observational period.
  Interventions: Drug: SerpinPC

INTERVENTIONS:
Drug: SerpinPC — Administered as SC injection.
  Other Names: Activated Protein C (APC) inhibitor

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, tolerability and pharmacokinetic (PK) profile of prophylactic SerpinPC in participants with Hemophilia B with inhibitors, as part of the SerpinPC registrational program.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants greater than or equal to (>=) 12 and less than or equal to (<=) 65 years of age at the time of informed consent.
2. Capable of providing written informed consent (adolescent assent and parental/guardian/legal representative consent when appropriate) for participation and having the opportunity to discuss the study with the Investigator or delegate.
3. Historically documented HemB (defined as factor IX <=0.05 international unit/Milliliter (IU/mL) [<=5 percent (%)]).
4. Participants who are currently in a prophylaxis program must be willing to stop prophylaxis (including episodic prophylaxis for sporting events) before the first dose of SerpinPC.
5. Historical or ongoing Factor IX inhibitor with bypass agents based on medical records or laboratory reports.
6. Documented ABR of 6 in the 12 months before screening (participants not on prophylaxis regimen) or documented ABR of ≥2 for participants on prophylaxis regimen
7. At least 12 weeks of prospective documentation of bleeding episodes in the AP-0105 (NCT05605678) non-interventional study before SerpinPC dosing, or willing to complete a 12-week observational period (at minimum) in AP-0103.
8. No bleeding in the 7 days before Baseline (the prospective observation period can be extended by 10 days if there is an ongoing active bleed).
9. D-dimer of <=750 micrograms/Liter (mc/L); in cases where there is a resolving bleed, the exclusion threshold is <=1750 mg/L at Screening and Pre-dosing visits.
10. Adequate hematologic function, defined as a platelet count of >=100,000/microliters (mcL) (>=100*10^9/L) and hemoglobin level of >=10 grams/deciliter(g/dL) (>=100 g/L or >= 6.206 millimoles per liter (mmol/L) at Screening and Pre-dosing visits.
11. Adequate hepatic function, defined as a total bilirubin level of <=1.5*upper limit of normal (ULN) (excluding Gilbert syndrome) and aspartate aminotransferase and/or alanine aminotransferase of <=3*ULN at Screening and Pre-dosing visits; no clinical signs or known laboratory or radiographic evidence consistent with cirrhosis of the liver.
12. Adequate renal function, defined as a serum creatinine level of <=2.0*ULN at Screening and Pre-dosing visits.
13. Able to use a diary to document bleeding events and medication usage.
14. Sexually active participants with a partner who could become pregnant should agree to use effective contraception for the duration of the study.

Effective contraceptive measure include condom with or without spermicide, a combination of male condom with either cap, diaphragm, or sponge with spermicide (double barrier methods), vasectomy, partner using stable contraceptive measures (combined [ estrogen and progestogen-containing] hormonal contraception or progestogen-only hormonal contraception initiated 2 or more menstrual cycles prior to screening, intrauterine device [IUD]. Intrauterine hormone-releasing system [IUS], bilateral tubal ligation), and/or sexual abstinence.

Exclusion Criteria:

1. Known severe thrombophilia (defined as antithrombin deficiency and/or protein S deficiency and/or protein C deficiency).
2. Participant with previous factor IX inhibitor who responded to immune tolerance induction and remains on prophylactic factor concentrate.
3. Previous deep vein thrombosis, pulmonary embolism, myocardial infarction, or stroke.
4. History of intolerance to SC injections.
5. Uncontrolled hypertension (systolic blood pressure >160 millimeter of mercury (mm Hg); diastolic blood pressure >100 mm Hg).
6. Weight >150 kilograms (kg) OR body mass index >40 kg/meter square (m^2).
7. Has active cancer and/or requires therapy for cancer, except for basal cell carcinoma.
8. Participation in another clinical trial (except for AP-0105 [NCT05605678]) during the 30 days before screening.
9. Prior, ongoing, or planned treatment with gene therapy for HemB
10. Any major medical, psychological, or psychiatric condition that could cause the participant to be unsuitable for the study or could interfere with the interpretation of the study results.
11. History of or other evidence of recent alcohol or drug abuse as determined by the Investigator (in the 12 months before screening).
12. Known human immunodeficiency virus (HIV) infection with CD4 count (or T-cell count) of <200 cells/mcL within 24 weeks before Screening and Pre-dosing visits. Patients with HIV infection who have CD4 > 200 and meet all other criteria are eligible.
13. Current or planned treatment with anticoagulant or antiplatelet drugs
14. Is planning to donate/bank sperm during SerpinPC treatment AND within 30 days of last dose of SerpinPC.
15. Any other significant conditions or comorbidities that, in the opinion of the Investigator, would make the participant unsuitable for enrollment, or could interfere with participation in, or completion of the study.

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Annualized Bleeding Rate (ABR) for Treated Bleeds up to Week 24 | Up to Week 24

SECONDARY OUTCOMES:
Annualized Bleeding Rate (ABR) for Treated Bleeds Up to Week 48 | Up to Week 48
Annualized Bleeding Rate (ABR) for Treated Spontaneous Bleeds | Up to Week 48
Annualized Bleeding Rate (ABR) for Treated Spontaneous Joint Bleeds | Up to Week 48
Total Coagulation Factor and/or Bypass Product Consumption During SerpinPC Treatment | Up to Week 48
Pharmacokinetic Concentrations of SerpinPC | From Day 1(Pre-dose) up to Week 48(Post-dose)
Haemophilia Quality-of-Life Questionnaire for Adults (Haem-A-QoL) Physical Health Scale | From Baseline up to Week 48
  The Haem-A-QoL instrument contains 44 items across 10 domains relevant to HRQoL in adults (physical health, feelings, view of participant's self, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, partnership, and sexuality). Each item is rated on a 5-point scale (1=never, 2=rarely, 3=sometimes, 4=often, 5=all the time). Higher scores are indicative of greater impairment in HRQoL.
Number of participants with Adverse events (AEs) | From Baseline up to Week 52
Number of Participants with Persistent High-titer Antidrug Antibodies (ADAs) | From Baseline up to Week 48
Number of Participants with Severity of Injection-site Reactions | Baseline up to Week 44

CONTACTS AND LOCATIONS:
Locations (20):
- United States (3):
  - University of Colorado School of Medicine, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - East Carolina University, Greenville, North Carolina
- Centre of Haematology named after prof. R. O. Yeolian/ Hemophilia center, Yerevan, Armenia
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- France (4):
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - CHRU de Lille Centre de biologie et pathologie, Lille
  - Hospices Civils de Lyon (HCL) - Hopital Femme-Mere-Enfant (HFME), Lyon
  - Hopital Necker - Enfants Malades, Paris
- University Hospital Frankfurt M, Frankfurt, Germany
- K J Somaiya Super Speciality Hospital & Research Centre, Mumbai, Maharashtra, India
- Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Italy
- Hospital Universitario La Paz, Madrid, Spain
- Taiwan (3):
  - Chung Shan Medical University, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
- Turkey (Türkiye) (2):
  - Istanbul University Oncology Institute, Istanbul
  - Ege University Medical Faculty Hospital, Izmir
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No